CLINICAL TRIAL: NCT01054079
Title: A Phase II Trial to Assess the Effect of Cinacalcet Hydrochloride on PSA Levels in Patients With Biochemically Recurrent Prostate Cancer After Failed Definitive Local Therapy
Brief Title: Cinacalcet Hydrochloride in Treating Men With Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00009741; NCI-2009-01514 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98309 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cinacalcet hydrochloride) (Experimental): Patients receive cinacalcet hydrochloride PO QD for 20 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: laboratory biomarker analysis; Procedure: quality-of-life assessment; Other: questionnaire administration; Drug: cinacalcet hydrochloride

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative study
Procedure: quality-of-life assessment — Ancillary study
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary study
Drug: cinacalcet hydrochloride — Given PO
  Other Names: Mimpara; Sensipar

SUMMARY:
This phase II trial is studying how well cinacalcet hydrochloride works in treating men with recurrent prostate cancer. Cinacalcet hydrochloride may be effective in lowering prostate-specific antigen (PSA) levels in patients with recurrent prostate cancer that has not responded to previous treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypothesis that once-daily treatment with 30 mg of cinacalcet hydrochloride (Sensipar) will reduce the rate of rise of serum prostate-specific antigen (PSA) compared to pre-treatment PSA values in subjects with biochemically recurrent prostate cancer after failed definitive local therapy.

OUTLINE:

Patients receive cinacalcet hydrochloride orally (PO) once daily (QD) for 20 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate
* For patients who have recurrent disease following surgery as first line therapy ("surgical failures")
* PSA requirement is 0.2 ng/ml or above
* For patients who have recurrent disease following radiation as first line therapy, the eligibility follows the "Phoenix criteria", that is, a rise of 2 ng/mL over the PSA nadir
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Granulocytes >= 1000/uL
* Serum creatinine =< 2.0 mg/dl
* Total serum calcium > 9.0 and < 10.5 mg/dl
* Total bilirubin =< 2.0 mg/dl
* Platelet count >=100,000/uL
* Hemoglobin (Hgb) >= 9 g/dL
* Total testosterone >= 50 ng/dL
* Ability to understand and the willingness to sign a written informed consent document (either directly or via a legally authorized representative)

Exclusion Criteria:

* Serious medical illness which would limit survival to less than 3 months
* Active, uncontrolled bacterial, viral or fungal infection
* Hemorrhagic disorder
* Any radiographic evidence of metastatic disease including positive bone scan or computed tomography (CT) abdomen/pelvis
* History of hypocalcemia or seizure disorder
* Patients with known hypersensitivity to any of the components of cinacalcet (cinacalcet hydrochloride)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K.C. Balaji, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Cinacalcet Hydrochloride)
Started | 20
# Recieved Proper PSA Testing | 10
Completed | 20 (while all 20 patients received at least some of the intervention, some did not get proper PSA tests.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cinacalcet Hydrochloride)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Rate of Rise of Serum PSA
Description: The difference of post treatment and pre-enrollment PSA.For those with multiple PSA measures post we use the median of those measures to estimate the participant's post PSA level.
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: Nanograms Per Milliliter
Arm/Group | Treatment (Cinacalcet Hydrochloride)
Number analyzed (Participants) | 10
Nanograms Per Milliliter | 0.0825 [-0.01 to 0.17]

2. Secondary Outcome: Change in Quality of Life (QOL) as Assessed by the Brief Male Sexual Inventory
Description: The Brief Male Sexual Inventory is an 11 question assessment including subscales: sex drive, erections, ejaculation. The scores are totaled to produce an overall score with a range of 1-45, with higher score indicating worse outcomes.
Time Frame: Up to 20 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment (Cinacalcet Hydrochloride)
Number analyzed (Participants) | 10
units on a scale
  baseline | 23.7 (2.7)
  20 weeks | 21.8 (2.2)

3. Secondary Outcome: Change in Hormonal Assessment Scale From Expanded Prostate Cancer Index Composite (EPIC)
Description: The Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. Epic produces two scores, one for function (5 items) and the other for bother (6 items). The response for each item is standardized to a 0 to 100 scale. For both scales, higher scores indicate worse outcomes.
Time Frame: up to 20 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment (Cinacalcet Hydrochloride)
Number analyzed (Participants) | 10
units on a scale
  baseline function | 86 (2.8)
  20 weeks function | 88 (3.1)
  baseline bother | 92.6 (1.6)
  20 weeks bother | 91.9 (1.6)

4. Secondary Outcome: Change in Functional Assessment of Cancer Therapy-Prostate (FACT-P)
Description: The FACT-P is a multidimensional, self-report QoL instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. Each item is rated on a 0 to 4 Likert type scale, and then combined to produce subscale scores for each domain, as well as a global QoL score. All subscale items are summed to a total. The score range is 0-156. Higher scores represent better quality of life.
Time Frame: up to 20 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment (Cinacalcet Hydrochloride)
Number analyzed (Participants) | 10
units on a scale
  baseline | 122.4 (3.4)
  20 weeks | 124.1 (3.1)

5. Secondary Outcome: Change in Total and Free Testosterone
Description: The detectable difference is estimated using a paired t-test approach. The lab measure will also be analyzed longitudinally using all measures with a mixed model approach adjusting for individual covariates.
Time Frame: Up to 20 weeks
Population: No data collected
Arm/Group | Treatment (Cinacalcet Hydrochloride)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Cinacalcet Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cinacalcet Hydrochloride) (N=20)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
hypocalcemia (Investigations) | 1 (1)
Hypoxia (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Lymphopenia (Investigations) | 1 (1)
Pulmonary hypertension (Cardiac disorders) | 1 (1)
Cardiac troponin T increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cinacalcet Hydrochloride) (N=20)
Nausea (Gastrointestinal disorders) | 2 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Neuropathy: sensory (Cardiac disorders) | 3 (3)
hypocalcemia (Investigations) | 14 (61)
hyponatremia (Investigations) | 1 (1)
Pruritus/itching (General disorders) | 1 (1)
Pain: Joint (General disorders) | 1 (4)
hypertriglyceridemia (Investigations) | 1 (1)
Pain: Muscle (General disorders) | 1 (1)
hypocalcemia (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes